CLINICAL TRIAL: NCT06033911
Title: A Randomized Controlled Trial Using FoodFlip©, a Mobile Phone App, to Promote Healthier Diets and Food Choices Among Post-Secondary Students
Brief Title: Using FoodFlip© to Improve Food Choices Among Post-secondary Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, Mary L'Abbe, Professor Emeritus, CM, PhD, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 508519; CIHR UD1-170157 (Other Grant/Funding Number: Canadian Institutes of Health Research)
Record Dates: First submitted 2023-09-05; First posted 2023-09-13 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Healthy Diet
Keywords: front-of-package labeling; post-secondary foods; university foods; universities; mobile applications; mobile health; smartphone

STUDY DESIGN:
Intervention Model Description: 2-week long, single-blinded randomized controlled trial with a 3-parallel arm.
Who Masked: Participant
Masking Description: Participants will be allocated into one of 3 groups: (i) no App control; (ii) App without 'high-in' nutrition symbol; (iii) App with Canada's 'high-in' nutrition symbol
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- No App (No Intervention): No intervention. Participants will be given access to a web-based submission portal.
- FoodFlip© App with no nutrition symbol (Placebo Comparator): Intervention control: participants will have access to food information in the shape of a Nutrition Facts table through FoodFlip©. Participants will have access to a submission portal linked to their study ID through the app.
  Interventions: Device: FoodFlip© App with no nutrition symbol
- FoodFlip© App with 'high-in' nutrition symbol (Active Comparator): Intervention: Participants will have access to food information through FoodFlip© with Health Canada's 'high-in' nutrition symbol. ©. Participants will have access to a submission portal linked to their study ID through the app.
  Interventions: Device: FoodFlip© App with 'high-in' nutrition symbol

INTERVENTIONS:
Device: FoodFlip© App with no nutrition symbol — Intervention control: participants will have access to food information such as calories or the Nutrition Facts table through FoodFlip©
  Arms: FoodFlip© App with no nutrition symbol
Device: FoodFlip© App with 'high-in' nutrition symbol — Intervention: Participants will have access to food information through FoodFlip© with Canada's 'high-in' NS
  Arms: FoodFlip© App with 'high-in' nutrition symbol

SUMMARY:
Canada passed mandatory front-of-package labelling (FOPL) regulations where pre-packaged food and beverage products that are high in sugar, saturated fat, and/or sodium are required to display a 'high-in' front-of-pack nutrition symbol (NS). FOPL is an effective tool to inform consumers about products that can harm health and help guide their purchasing decisions. However, as the regulations are limited to the pre-packaged food supply and do not apply to restaurants and other food services, little is known about the potential impact of the NS in such settings. Therefore, the objective of the present study is to investigate the impact of the Canadian FOPL (i.e. the 'high-in' NS) as delivered through a mobile health (mHealth) app in a setting currently not subject to regulations. The study will take place on a post-secondary campus (University of Toronto) hosting students, a population vulnerable to poor dietary choices, nutritional knowledge, and associated weight gain. A 2-week long, randomized controlled trial with a 3-parallel arm study design will be conducted to explore the effect of the 'high-in' NS on students' purchasing behaviours and nutritional knowledge. Eligible participants will be randomly allocated into one of 3 intervention groups: no App control; App control with no NS; App with NS. Questionnaires will be used to assess nutritional knowledge, and receipts will be used to analyze purchasing behaviour.

DETAILED DESCRIPTION:
Poor diets increase the risk of non-communicable diseases (NCDs), one of the major causes of disability and premature mortality in Canada. To help improve the diets of Canadians, Health Canada recently promulgated front-of-pack labelling (FOPL) regulations, which mandate pre-packaged foods and beverages meeting and/or exceeding the thresholds for nutrients of public health concern (i.e., sugars, saturated fat, and/or sodium) to display a 'high-in' front-of-pack nutrition symbol (NS). Moreover, previous studies have shown that FOPL can improve purchasing behaviours of consumers by decreasing purchases of nutrients of public health concern and/or foods carrying 'less healthy' FOPL and increase the nutritional knowledge of consumers. However, the FOPL regulations do not address restaurant foods, which are significant caloric contributors to the Canadian diet and are often high in nutrients of public health concern. Further, FOPL regulations do not address foods sold in other institutional settings, including schools, long-term care homes, and daycares. This policy gap may adversely affect the young adult population - a group notably vulnerable to poor diets and associated weight gain and poor nutritional knowledge. Emerging evidence suggests that FOPL can be an effective tool to communicate nutrition information to promote healthier food choices in food service settings; however, limited data exist on the effectiveness of FOPL on menu items available on post-secondary campuses to influence students' food purchasing behaviours on campus and to improve their nutritional knowledge. Furthermore, nutrition mobile health (mHealth) apps have been shown to have the potential to support behavioural change, improve nutrition knowledge, and develop skills to promote healthy eating behaviours through quick information-sharing capacity, customizable tracking abilities, and interactive components. The L'Abbe Lab has developed a mobile application, FoodFlip©, that provides nutrition information at the point of purchase to influence the decision-making process with high usability and functionality in grocery shopping settings. However, the application of FoodFlip© on purchasing behaviours in post-secondary campus settings is unknown. Therefore, the primary objective of the study is to investigate the effect of the Canadian FOPL (i.e., the 'high-in' nutrition symbol) on purchasing behaviours and nutritional knowledge of post-secondary students on campus, using the FoodFlip© App.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* enrolled at UofT
* have regular access to either iPhone or Android
* purchases at least one meal a day on campus
* able to speak and read English
* not currently pregnant or in lactation

Exclusion Criteria:

* <18 years of age
* not enrolled at UofT
* does not have access to a smartphone
* does not purchase at least one meal a day on campus
* unable to speak and read English
* currently pregnant or in lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2024-01-29 (Actual); Primary Completion 2024-04-22 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Purchasing Behaviors | 2 weeks
  Purchasing behaviours will be assessed using receipts and/or records provided by participants over the 2-week study period. Nutritional quality of purchased menu items will be determined using a nutrient profiling model based on the thresholds for Canada's FOPL regulations. Menu items will be assigned a "Menu item score" on a scale of 0 (minimum) to 3 (maximum), with 0 indicating no 'high-in' nutrients and 3 being 'high-in' all 3 nutrients-of-concern. Scores of each menu item purchased will be summed and divided by the total number of purchases to derive the final score for each participant; higher scores mean lower nutritional quality (i.e. worse outcome) and lower scores mean higher nutritional quality (i.e. better outcome). The final scores will then be compared between intervention groups, and change in nutritional quality will be compared within intervention groups at 2 time points: early intervention (end of Week 1) and late intervention (end of study period).
Nutritional Knowledge | 2 weeks
  Nutritional knowledge will be assessed using an online questionnaire developed and validated by the L'Abbe Lab. Questionnaire will be completed by participants at 1) baseline and 2) end-of-study. This short (10-15 min) survey of 30 short questions will include questions assessing health literacy and nutritional knowledge that have been adapted from validated questionnaires. Correct answers will be coded as "1" while incorrect answers will be coded as "0", with a maximum of 30 points. Higher scores indicate higher nutritional knowledge (i.e. better outcome), and lower scores indicate lower nutritional knowledge (i.e. worse outcome). Between intervention groups differences in nutritional knowledge will be assessed using ANOVA, while changes in nutritional knowledge from baseline to end-of-study will be compared within intervention groups using Mann-Whitney U-tests.

CONTACTS AND LOCATIONS:
Overall Officials: Mary R L'Abbe, PhD, Principal Investigator — University of Toronto; Hayun Jeong, HBSc, Study Director — University of Toronto
Locations (1):
- Department of Nutritional Sciences, University of Toronto, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] World Health Organization, Chronic diseases and their common risk factors. 2005 [cited 2021 Sept 1]; Available from: https://www.who.int/chp/ chronic_disease_report/media/Factsheet1.pdf.
- [Background] World Health Organization, Noncommunicable diseases country profiles 2018. 2018 [cited 2021 Sept 1]; Available from: https://www.who.int/nmh/ publications/ncd-profiles-2018/en/.
- [Background] Health Canada. Regulations Amending the Food and Drug Regulations (Nutrition Symbols, Other Labelling Provisions, Vitamin D and Hydrogenated Fats or Oils) [Internet]. Canada Gazette, Part II. 2022. Available from: https://canadagazette.gc.ca/rp-pr/p2/2022/2022-07-20/html/sor-dors168-eng.htmlHealth.
- [Background] Vergeer L, Vanderlee L, Ahmed M, Franco-Arellano B, Mulligan C, Dickinson K, L'Abbe MR. A comparison of the nutritional quality of products offered by the top packaged food and beverage companies in Canada. BMC Public Health. 2020 May 11;20(1):650. doi: 10.1186/s12889-020-08828-w. PMID 32393206
- [Background] Ang FJL, Agrawal S, Finkelstein EA. Pilot randomized controlled trial testing the influence of front-of-pack sugar warning labels on food demand. BMC Public Health. 2019 Feb 7;19(1):164. doi: 10.1186/s12889-019-6496-8. PMID 30732609
- [Background] Neal B, Crino M, Dunford E, Gao A, Greenland R, Li N, Ngai J, Ni Mhurchu C, Pettigrew S, Sacks G, Webster J, Wu JH. Effects of Different Types of Front-of-Pack Labelling Information on the Healthiness of Food Purchases-A Randomised Controlled Trial. Nutrients. 2017 Nov 24;9(12):1284. doi: 10.3390/nu9121284. PMID 29186803
- [Background] Taillie LS, Reyes M, Colchero MA, Popkin B, Corvalan C. An evaluation of Chile's Law of Food Labeling and Advertising on sugar-sweetened beverage purchases from 2015 to 2017: A before-and-after study. PLoS Med. 2020 Feb 11;17(2):e1003015. doi: 10.1371/journal.pmed.1003015. eCollection 2020 Feb. PMID 32045424
- [Background] Vanderlee L, Franco-Arellano B, Ahmed M, Oh A, Lou W, L'Abbe MR. The efficacy of 'high in' warning labels, health star and traffic light front-of-package labelling: an online randomised control trial. Public Health Nutr. 2021 Jan;24(1):62-74. doi: 10.1017/S1368980020003213. Epub 2020 Oct 6. PMID 33019950
- [Background] Statistics Canada Eating out - How often and why [Stats in brief: 11-627-M2019003], Statistics Canada: Ottawa, Ontario. 2019.
- [Background] Moubarac, J.C., Ultra-processed foods in Canada: consumption, impact on diet quality and policy implications. University of Montreal: Montreal. 2017.
- [Background] Yang Y, Weippert M, Ahmed M, L'Abbe MR. Cross-Sectional Nutritional Information and Quality of Canadian Chain Restaurant Menu Items in 2020. Am J Prev Med. 2023 Jan;64(1):42-50. doi: 10.1016/j.amepre.2022.07.015. Epub 2022 Sep 22. PMID 36155709
- [Background] Murphy SA, Weippert MV, Dickinson KM, Scourboutakos MJ, L'Abbe MR. Cross-Sectional Analysis of Calories and Nutrients of Concern in Canadian Chain Restaurant Menu Items in 2016. Am J Prev Med. 2020 Oct;59(4):e149-e159. doi: 10.1016/j.amepre.2020.05.005. Epub 2020 Aug 20. PMID 32828587
- [Background] Vella-Zarb RA, Elgar FJ. The 'freshman 5': a meta-analysis of weight gain in the freshman year of college. J Am Coll Health. 2009 Sep-Oct;58(2):161-6. doi: 10.1080/07448480903221392. PMID 19892653
- [Background] Levitsky DA, Halbmaier CA, Mrdjenovic G. The freshman weight gain: a model for the study of the epidemic of obesity. Int J Obes Relat Metab Disord. 2004 Nov;28(11):1435-42. doi: 10.1038/sj.ijo.0802776. PMID 15365585
- [Background] Matthews JI, Doerr L, Dworatzek PDN. University Students Intend to Eat Better but Lack Coping Self-Efficacy and Knowledge of Dietary Recommendations. J Nutr Educ Behav. 2016 Jan;48(1):12-19.e1. doi: 10.1016/j.jneb.2015.08.005. Epub 2015 Sep 28. PMID 26424531
- [Background] Block JP, Roberto CA. Potential benefits of calorie labeling in restaurants. JAMA. 2014 Sep 3;312(9):887-8. doi: 10.1001/jama.2014.9239. No abstract available. PMID 25077460
- [Background] West JH, Belvedere LM, Andreasen R, Frandsen C, Hall PC, Crookston BT. Controlling Your "App"etite: How Diet and Nutrition-Related Mobile Apps Lead to Behavior Change. JMIR Mhealth Uhealth. 2017 Jul 10;5(7):e95. doi: 10.2196/mhealth.7410. PMID 28694241
- [Background] McCarroll R, Eyles H, Ni Mhurchu C. Effectiveness of mobile health (mHealth) interventions for promoting healthy eating in adults: A systematic review. Prev Med. 2017 Dec;105:156-168. doi: 10.1016/j.ypmed.2017.08.022. Epub 2017 Sep 4. PMID 28882743
- [Background] Ahmed M, Oh A, Vanderlee L, Franco-Arellano B, Schermel A, Lou W, L'Abbe MR. A randomized controlled trial examining consumers' perceptions and opinions on using different versions of a FoodFlip(c) smartphone application for delivery of nutrition information. Int J Behav Nutr Phys Act. 2020 Feb 12;17(1):22. doi: 10.1186/s12966-020-0923-1. PMID 32050996
- [Background] Pan American Health Organization. Front-of-package labeling [Internet]. Available from: https://www.paho.org/en/topics/front-package-labeling